CLINICAL TRIAL: NCT02138669
Title: INTACS® Prescription Inserts Used to Treat Patients With Keratoconus as a Humanitarian Use Device
Brief Title: Intacs Prescription Inserts for Keratoconus Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Steven Verity, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 012011-115; Intacs_Prospective (Other: UTSW - Department of Ophthalmology)
Record Dates: First submitted 2014-05-05; First posted 2014-05-14 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Keratoconus
Keywords: Cornea; Keratoconus; Steep cornea
MeSH Terms: conditions — Keratoconus; Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Intacs Device (Other): INTACS® prescription inserts are an ophthalmic medical device designed for the reduction or elimination of myopia and astigmatism in patients with keratoconus so that their functional vision may be restored and the need for a corneal transplant procedure can potentially be deferred.
  Interventions: Device: Intacs

INTERVENTIONS:
Device: Intacs — INTACS® prescription inserts are an ophthalmic medical device designed for the reduction or elimination of myopia and astigmatism in patients with keratoconus so that their functional vision may be restored and the need for a corneal transplant procedure can potentially be deferred.

SUMMARY:
The US food and Drug Administration (FDA) originally approved INTACS prescription inserts in April 1999 for the correction of low levels of nearsightedness (-1.00 to -3.00 diopters). Additional clinical data have shown that INTACS are safe for the treatment of keratoconus, in July 2004, FDA approved INTACS inserts for the treatment of keratoconus as a Humanitarian Use Device (FDA approval letter attached). The statute and the implementing regulation of FDA (21 CFR 814.124 (aj) require IRB review and approval before a HUD is used.INTACS prescription inserts are composed of two clear segments, each having an arc length of 150°, they are manufactured form a biomedical material called polymethylmethacrylate (PMMA) and are available in three thicknesses. Two INTACS inserts ranging from 0.250mm to 0.350mm may be implanted depending on the orientation of the cone and the amount of myopia and astigmatism to be reduced.

DETAILED DESCRIPTION:
The INTACS procedure is typically performed in an outpatient setting. The two tiny INTACS inserts are surgically placed into the periphery of the cornea through a tiny cut that is made on the cornea after numbing drops have been applied. A specially designed instrument creates a tunnel by separating the tissue layers in the outside periphery of the cornea, the INTACS inserts are placed into this tunnel where they remain. One or two ophthalmic sutures will be placed to close the incision. A postoperative care information booklet will be given to the patients; patients will be followed by means of postoperative appointments for up to 12 months after the surgery. The visits/testing schedules are listed below:

Pre-OR visit (1.5 hours): Visual Acuity (VA), Refraction, Topography, Keratometry, Glare Test. Mesopic Pupil Size, Pachymetry, Tonometry, Slit Lamp Exam and Contrast Sensitivity.

Surgery (30min): At Laser Center for Vision Care which is part of Aston and department of Ophthalmology.

Post-OR Day 1(10min): VA, Slit Lamp Exam.

Post-OR 1week (20min): Visual Acuity, Refraction, Topography, Tonometry, Slit Lamp Exam.

Post-OR 1 month (20minj: Visual Acuity, Refraction, Topography, Tonometry, Slit Lamp Exam.

Post-OR 3 month (1.5 hours): Some as pre-op Visit.

Post-OR 6 month (20min): Visual Acuity, Refraction, Topography, Tonometry, Slit Lamp Exam.

Post-OR 12 month (1.5 hours): Same as pre-op.

ELIGIBILITY:
Inclusion Criteria:

Who have experienced a progressive deterioration in their vision, such thot they can no longer achieve adequate functional vision on a daily basis with their contact lenses or spectacles; Who are 21 years of age or older; Who have clear central corneas; Who have a corneal thickness of 450 microns or greater at the proposed incision site; Who have corneal transplantation as the only remaining option to improve their functional vision.

Exclusion Criteria:

Who have abnormally thin corneas or who have a corneal thickness of 449 microns or less at the proposed incision site;

Patients with collagen vascular, autoimmune or immunodeficiency disease;

Pregnant or nursing patients;

Presence of ocular conditions, such as recurrent corneal erosion syndrome or corneal dystrophy, that my predispose the patient to future complications;

Patients who are taking on or more of following medications: isotretinoin (Accutane); amiodarone HCL (Cordarone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-01; Primary Completion 2027-12-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of INTACS prescription inserts to reduce astigmatism due to Keratoconus as determined by refraction assessment. | 12 Months
  INTACS® prescription inserts are used to treat patients with Keratoconus as a Humanitarian Use Device. Efficacy of the INTACS inserts to reduce the effects of Keratoconus will be assessed using Refraction (pre-op refraction will be evaluated post-operatively) to assess the effectiveness of INTACS surgery in regards decreasing level of astigmatism.
Efficacy of INTACS prescription inserts to reduce astigmatism due to Keratoconus as determined by visual acuity examination. | 12 Months
  INTACS® prescription inserts are used to treat patients with Keratoconus as a Humanitarian Use Device. Efficacy of the INTACS inserts to reduce the effects of Keratoconus will be assessed using Visual Acuity to assess the effectiveness of INTACS surgery in regards decreasing level of astigmatism.
Efficacy of INTACS prescription inserts to reduce other corneal aberrations due to Keratoconus as determined by corneal topography assessment. | 12 Months
  Corneal Topography evaluation to assess post-operative vs. pre-operative corneal surface curvature differences will be used to measure efficacy of this INTACS prescription inserts, and an evaluation whether there is a need for further interventions, including corneal transplant.
Efficacy of INTACS prescription inserts to reduce other corneal aberrations due to Keratoconus as determined by tonometry assessment. | 12 Months
  Tonometry will be used to measure efficacy of this INTACS prescription inserts, and an evaluation whether there is a need for further interventions, including corneal transplant.
Efficacy of INTACS prescription inserts to reduce other corneal aberrations due to Keratoconus as determined by slit lamp corneal examination. | 12 Months
  Slit Lamp corneal examination will be used to measure efficacy of this INTACS prescription, and an evaluation whether there is a need for further interventions, including corneal transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Verity, MD, Principal Investigator — UTSW Medical Center at Dallas
Locations (1):
- UTSW Medical Center at Dallas, Dallas, Texas, United States